CLINICAL TRIAL: NCT02429869
Title: Impact of Everolimus on HIV Persistence Post Kidney (and Kidney/Pancreas) or Liver Transplant
Brief Title: Impact of Everolimus on HIV Persistence Post Kidney or Liver Transplant
Acronym: HIVTR-EVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: amfAR, The Foundation for AIDS Research (Other); Novartis (Industry)
Responsible Party: Principal Investigator, Peter Stock, Professor of Surgery, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HIVTR-EVE
Record Dates: First submitted 2015-04-24; First posted 2015-04-29 (Estimated); Results first posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-10

CONDITIONS: HIV; Kidney Transplant; Liver Transplant
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus (Experimental)
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus
  Other Names: Zortress

SUMMARY:
Zortress (everolimus), the 40-O-(2-hydroxyethyl)-derivative of rapamycin, is an mTOR inhibitor approved for rejection prophylaxis in kidney transplant recipients. mTOR inhibition may favorably impact the HIV viral reservoir, and we hypothesize that adding everolimus to the transplant immunosuppressive regimen of HIV positive transplant recipients will decrease HIV persistence in CD4+ lymphocytes.

DETAILED DESCRIPTION:
Open-label, single arm study that will enroll antiretroviral-treated HIV-infected adults who are doing well post-liver or post-kidney transplant who are eligible and willing to add everolimus to their immunosuppressive regimen (with a target trough level between 3-8 ng/ml). Calcineurin inhibitors will be decreased to obtain a 50% reduction in trough levels with the addition of everolimus. Subjects will be maintained on that regimen for 6 months.

Biologic specimens for intensive immunology and virology studies will be obtained before, during and after exposure to everolimus. Samples will be analyzed at screening, baseline (prior to addition of everolimus), and at weeks 8 and 26 (while on everolimus), and week 52 (6 months post everolimus discontinuation).

ELIGIBILITY:
Inclusion Criteria:

1. Solid organ (kidney, kidney/pancreas, or liver) transplant recipient
2. Male or female ≥ 18 years of age.
3. Documentation of HIV-1 infection diagnosis as evidenced by any licensed ELISA and confirmation by Western Blot, or documented history of detectable HIV-1 RNA)
4. HIV-1 plasma RNA <50 copies/ml for at least 2 years with at least one measurement per year and most recent viral load within 16 weeks of enrollment and study drug initiation. Episodes of a single HIV plasma RNA 50 - 500 copies/ml will not exclude participation if the subsequent HIV plasma RNA was <50 copies/ml.
5. CD4+ T cell counts greater than 200 cell/µl within 16 weeks of enrollment and study drug initiation.
6. Receiving combination antiretroviral therapy (at least 3 agents)
7. Written informed consent obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
3. Patients who are intending to modify antiretroviral therapy in the next 6 months for any reason.
4. Serious illness requiring hospitalization or parenteral antibiotics within preceding 3 months.
5. A screening hemoglobin below 11.5 g/dL.
6. A screening TSH consistent with hypothyroidism.
7. Significant renal disease (eGFR < 60 ml/min) or acute nephritis
8. Clinically active hepatitis as evidenced by clinical jaundice or Grade 2 or higher liver function test abnormalities.
9. Hepatic cirrhosis or decompensated chronic liver disease.
10. Concurrent treatment with immunomodulatory drugs, such an interferon-alpha, or exposure to any immunomodulatory drug in past 16 weeks (outside of standard immunosuppression).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Henrich TJ, Schreiner C, Cameron C, Hogan LE, Richardson B, Rutishauser RL, Deitchman AN, Chu S, Rogers R, Thanh C, Gibson EA, Zarinsefat A, Bakkour S, Aweeka F, Busch MP, Liegler T, Baker C, Milush J, Deeks SG, Stock PG. Everolimus, an mTORC1/2 inhibitor, in ART-suppressed individuals who received solid organ transplantation: A prospective study. Am J Transplant. 2021 May;21(5):1765-1779. doi: 10.1111/ajt.16244. Epub 2020 Sep 15. PMID 32780519

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten HIV-infected adult solid organ transplant participants on stable ART and were taking non-mTOR based immune suppressive regimens for allograft rejection were recruited at the University of California, San Francisco in this open label, single-arm everolimus trial.
Groups:
- Everolimus: Subjects on mTOR inhibitor (everolimus) for 6 months, added to standard of care immunosuppressive regimen
Period: Overall Study
Arm/Group | Everolimus
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 58.5 [48 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Cell-associated HIV DNA
Description: Peripheral blood mononuclear cells were isolated from whole blood using the Ficoll density gradient technique. Peripheral blood CD4 T cells were enriched by negative selection using antibody-coupled magnetic beads (Stem Cell Technologies) prior to simultaneous RNA and DNA isolation using cell-sparing protocols (AllPrep, Qiagen). Bulk CD4+ T cell or PBMC-associated HIV DNA and unspliced RNA were quantified using real-time PCR methods.The primer and probe sequences targeted conserved regions to enable quantification of a broad range of HIV subtypes. Values were normalized to DNA quantification of a human housekeeping gene (CCR5) in order to determine nucleic acid copies per million CD4+ T cell or PBMC as described. In addition to traditional quantitative PCR, a novel single-cell-in-droplet (scd)PCR method was used to quantify the absolute number or frequency of individual purified CD4+ T cells that express unspliced HIV RNA.
Time Frame: Baseline, Month 2, Month 6, Month 12 (6 months post discontinuation of everolimus)
Population: CD4+ T Cell count was not collected at Month 6 for one participant who did not show up for the visit.
Measure: Median (Inter-Quartile Range); unit: nucleic acid copies per million cells
Groups:
- Everolimus: This is a single arm study. Subjects on mTOR inhibitor (everolimus) for 6 months, added to standard of care immunosuppressive regimen
Arm/Group | Everolimus
Number analyzed (Participants) | 10
nucleic acid copies per million cells
  Baseline | 35 [8 to 173]
  Month 2 | 43 [21 to 417]
  Month 6: number analyzed (Participants) | 9
  Month 6 | 81 [28 to 210]
  Month 12 | 16 [9 to 804]

2. Secondary Outcome: Cell-associated Total HIV RNA
Description: as for outcome 1
Time Frame: Baseline, Month 2, Month 6, Month 12 (6 months post discontinuation of everolimus)
Population: CD4+ T Cell count was not collected at Month 6 for one participant who did not show up for the visit.
Measure: Median (Inter-Quartile Range); unit: nucleic acid copies per million cells
Arm/Group | Everolimus
Number analyzed (Participants) | 10
nucleic acid copies per million cells
  Baseline HIV RNA CD4+ | 423 [148 to 1702]
  Month 2 HIV RNA CD4+ | 310 [228 to 789]
  Month 6 HIV RNA CD4+: number analyzed (Participants) | 9
  Month 6 HIV RNA CD4+ | 702 [417 to 1299]
  Month 12 HIV RNA CD4+ | 354 [165 to 633]

3. Secondary Outcome: Plasma HIV RNA
Description: Plasma HIV RNA was quantified in a highly sensitive single-copy assay (SCA) using repetitive sampling in the Panther system (Hologic) at the Blood Systems Research Institute. Up to 18 replicates were tested for each sample in order to determine plasma RNA levels as low as 0.18 copies/mL.
Time Frame: Baseline, Month 2, Month 6, Month 12 (6 months post discontinuation of everolimus)
Population: CD4+ T Cell count was not collected at Month 6 for one participant who did not show up for the visit.
Measure: Median (Inter-Quartile Range); unit: nucleic acid copies per million cells
Arm/Group | Everolimus
Number analyzed (Participants) | 10
nucleic acid copies per million cells
  Baseline | 0.291 [0 to 0.9283]
  Month 2 | 0.584 [0 to 1.547]
  Month 6: number analyzed (Participants) | 9
  Month 6 | 1.042 [0.189 to 2.05]
  Month 12 | 0.941 [0.191 to 1.576]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Everolimus
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus (N=10)
Gastritis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study had several obvious limitations, such as concomitant use of other immunomodulatory medications that may have masked or altered the effects of mTOR inhibition on HIV persistence. Sample size was also limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT02429869/Prot_SAP_000.pdf